CLINICAL TRIAL: NCT05018026
Title: A Randomized Trial and Impact Evaluation of Singapore's New Food Labels Aimed to Address the War on Diabetes
Brief Title: Understanding Grocery Shopping Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Soye Shin, Research Fellow, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Duke-NUS-KPFA/2020/0042
Record Dates: First submitted 2021-08-13; First posted 2021-08-24 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Diet Quality
Keywords: Nutri-Grade labels; Diet quality; Sugar-sweetened beverages; Online grocery shopping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Control Arm) (No Intervention): A default NUSMart that mirrors a conventional web-grocery store in Singapore where some healthier products are displayed with Singapore's Healthier Choice Symbol (HCS) logos (Control).
- Arm 2 (Nutri-Grade Arm) (Experimental): Similar to Arm 1 except that beverages will be displayed with a color-coded and graded Nutri-Grade label.
  Interventions: Behavioral: Nutri-Grade labels

INTERVENTIONS:
Behavioral: Nutri-Grade labels — All beverage products in the arm are displayed with the Nutri-Grade label. This label was proposed by the Ministry of Health in Singapore to be implemented at the end of 2021. It will apply to all pre-packaged non-alcoholic beverages sold in Singapore. It will have four color-coded grades wherein Grade A, corresponding to the lowest sugar and saturated fat thresholds, will be in green and Grade D, corresponding to the highest sugar and saturated fat thresholds, will be in red.
  Arms: Arm 2 (Nutri-Grade Arm)

SUMMARY:
This study aims to systematically evaluate the effect of Singapore's new front-of-pack non-alcoholic beverage labels, called Nutri-Grade, on the consumption of processed beverages. Using a fully functional grocery webstore, the investigators wish to assess the causal effect of the new labels on food and beverage purchase, sugar intake, and overall diet quality and examine how this effect varies by shoppers' income and education level.

The investigators' hypotheses about the effects of these new food labels, measured by the grams of sugar per serving (primary) of finalized shopping baskets, are as follows:

1. Hypotheses 1: The new sugar-sweetened beverage (SSB) labels will shift consumers toward healthier products. Sugar-sweetened beverages are any liquids that have been sweetened with one or more of the different forms of added sugars.
2. Hypotheses 2: The new SSB labels will reduce overall sugar and calories purchased and increase overall diet quality.
3. Hypotheses 3: Effects will be greater for those with low income/low education as they are least familiar with the nutrition facts panel and thus most likely to benefit from the new information.

DETAILED DESCRIPTION:
1. Experimental Design and Procedures

   The aim of this study is to use a 2 x 2 within-subject crossover design with an online grocery store, to systematically evaluate the effect of the new SSB front-of-pack labels, Nutri-Grade, on diet quality and examine how this effect varies by shoppers' income and education level. To this end, the investigators will be using two different versions of an online experimental grocery store called NUSMart, designed for research purposes. The two versions are described below.
2. Overview of Experimental Design

The investigators will recruit Singapore residents aged 21 years or older. Prospective participants will be asked to complete an online screener to determine their eligibility to participate in the study. Those who do not consent or are deemed ineligible will be notified of their ineligibility with an on-screen message.

If interested and eligible, the applicant will then be asked to complete a registration form containing name, mobile number, and email address. Contact information for the Duke-NUS study team will be provided to allow questions to be asked at any point in the consent process and throughout the study. Upon completion of the registration form, NUSMart will create the participant account and a unique ID number (CID) for use throughout the study. Participants will receive an automated email with their unique login details.

Participants will be directed to read the Participant Information Sheet and provide consent. The investigators will provide information on study protocols and participation details without disclosing the intervention arms explicitly, to maintain the integrity of participant responses and hence to ensure validity of results. It will be deleterious to the study to reveal the labels or the differences between study arms before participants complete both shops as this will likely confound participant responses. The consent form will state that in each of the shops there is a 50% chance that the participant will have to make actual purchases i.e. buy the groceries in the cart they checked out. In reality, it will be randomly decided earlier whether shopping trip 1 or 2 is the real shop. This will be achieved via a collaboration with a local online grocery provider, FairPrice.

After obtaining consent, participants will be asked to fill in a baseline survey to collect demographic and health characteristics. The baseline questionnaire includes a question as to whether any household members have a medical condition, such as diabetes or hypertension, which requires limiting the types of foods they eat.

Eligible participants who have completed to this point will enter a participant waiting list, where the study team will manually enroll the participant as active according to the capacity of the study team. Once participants have successfully enrolled in the study they will be informed by email, and are expected to complete two grocery shops (one shop per week) on NUSMart. Participants are expected to complete one shop in one sitting. The investigators will apply a within person design and randomize the order of the two shops. Participants will receive email and text reminders each week to complete their order.

Each participant will be told that they must buy at least one beverage product and that they will make the payment using their credit card & receive their grocery orders. This real-shopping experiment ensures the credibility of the results. Each participant will therefore shop a total of 2 times during the study. This will include 1 shop within each shopping condition (Arm 1 and Arm 2).

During the study, participants will be asked to purchase their weekly groceries the amount of which is similar to their typical grocery shopping for their households, with a specified minimum spend at each shop. A wheel of purchase will be used to determine which one of the 2 shops will the participant actually pay for and receive ordered goods for. Upon completion of their second shop, participants will be asked to fill in a short post-study survey asking for their feedback on the interventions. Participants who successfully complete both shops and all other surveys will be considered as having completed the study. Participants will be provided with the debriefing sheet via email after study completion. For the participants who wish to withdraw midway into the study, the debriefing sheet will be sent to them as soon as possible after they withdraw.

ELIGIBILITY:
Inclusion Criteria:

* Singapore resident
* Age 21 and above
* Must be the primary weekly grocery shopper in their household
* Must have an account with our appointed online grocery service provider or is willing to create one.

Exclusion Criteria:

* Non-Singapore resident
* Non-primary grocery shopper in their household
* Less than 21 years old
* Doesn't have an account with our appointed online grocery service provider and is unwilling to create one.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Sugar Levels | After completion of data collection, an average of about 5 months
  Grams of sugar per serving

SECONDARY OUTCOMES:
Calorie Intake | After completion of data collection, an average of about 5 months
  Calorie intake per serving and per shopping trip (kcal)
Purchased Beverage Quality | After completion of data collection, an average of about 5 months
  The proportion of Nutri-Graded C and D beverage servings purchased
Overall Diet Quality | After completion of data collection, an average of about 5 months
  Overall diet quality as measured by the average Nutri-Score weighted by the number of serving size. Nutri-Score is an individual dietary index based on the British Food Standard Agency Nutrient Profiling System.

CONTACTS AND LOCATIONS:
Overall Officials: Soye Shin, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin S, Puri J, Finkelstein E. A randomized trial to evaluate the impact of Singapore's forthcoming Nutri-grade front-of-pack beverage label on food and beverage purchases. Int J Behav Nutr Phys Act. 2023 Feb 15;20(1):18. doi: 10.1186/s12966-023-01422-4. PMID 36793058